CLINICAL TRIAL: NCT04966312
Title: Instructor School of Nursing, Chung Shan Medical University, Taichung, Taiwan
Brief Title: Preoperative Educational Videos Reduce Maternal Anxiety Whose Children Received Congenital Heart Disease Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University Hospital (Other)
Responsible Party: Sponsor-Investigator, Chung Shan Medical University Hospital, Department of pediatrics, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CS13143
Record Dates: First submitted 2021-06-07; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Educational Videos; Maternal Anxiety; Surgery; Congenital Heart Disease in Children; Maternal Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): mothers receiving routine education plus digital video disk before surgery
  Interventions: Other: Preoperative educational videos plus routine education
- control group (Other): mothers receiving routine education
  Interventions: Other: Preoperative routine education

INTERVENTIONS:
Other: Preoperative educational videos plus routine education — Mothers receiving routine education plus digital video disk before their children receiving congenital heart disease surgery. The content was the same as the routine education but was presented audio-visually, and the video was easy to understand by the general public.
  Arms: study group
Other: Preoperative routine education — Mothers receiving routine education before their children receiving congenital heart disease surgery
  Arms: control group

SUMMARY:
To examine if educational digital video disk can reduce maternal anxiety and depression if their children undergo congenital heart disease surgery and when surgical or post-surgical complications occur. Compared to only routine education, adding digital video disk could decrease mothers' anxiety more after education, and until the day of discharge. Compared to only routine education, adding digital video disk could decrease mothers' anxiety more on the discharge day if their child had surgical or post-surgical complications.

DETAILED DESCRIPTION:
Aims and objectives: To examine if educational digital video disk can reduce maternal anxiety and depression if their children undergo congenital heart disease surgery and when surgical or post-surgical complications occur.

Background: Mothers experience anxiety and depression if their children undergo conditions mentioned above.

Design: A randomized control-group pretest-posttest design. The CONSORT checklist is used.

Methods: In a teaching hospital, 120 mothers whose children underwent first elective surgery for congenital heart disease were randomly divided into group 1: 60 mothers receiving routine education plus digital video disk before surgery; and group 2: 60 mothers receiving routine education. Between groups, mothers' anxiety and depression levels were compared (1) before education, (2) after education (before surgery) and (3) on the discharge day. Among mothers whose children had surgical or post-surgical complications, the effect of watching the digital video disk on anxiety and depression at discharge day was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Mothers, whose children underwent first elective cardiac surgery for congenital heart disease
* Mothers should have been the primary caregivers
* Mothers able to communicate effectively, either orally or in writing

Exclusion Criteria:

* Mothers of children with genetic disorders
* Mothers of children with non-cardiac congenital anomalies
* Mothers of children with diseases such as cerebral palsy, epilepsy, psychiatric diseases, and * * Mothers of children with chronic lung diseases

Ages: 23 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of Mother's anxiety | day 1 (baseline, before education), day 1 (after education), day 5-7 (discharge day)
  The number scores of mother's anxiety between "routine education" and "routine plus DVD education" groups.
  Beck Anxiety Inventory (BAI) was used to evaluate the number scores of anxiety.
The change of Mother's depression | day 1 (baseline, before education), day 1 (after education), day 5-7 (discharge day)
  The number scores of mother's depression between "routine education" and "routine plus DVD education" groups.
  Beck Depression Inventory (BDI) was used to evaluate the number scores of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan